CLINICAL TRIAL: NCT00515138
Title: A Pilot Study of Standard-Dose Rituximab, Ifosfamide, Carboplatin and Etoposide (RICE) Plus Bortezomib (Velcade) in a Dose-Escalating Fashion for Patients With Relapsed or Primary Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma Who Are Candidates for Autologous Stem Cell Transplant
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator left institution. 7 patients accrued and there is insufficient data to analyze.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-CC06253
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Lymphoma, B-Cell
Keywords: B-Cell NHL; Autologous Stem Cell Transplant; RICE
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab; Ifosfamide; Carboplatin; Etoposide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab, Ifosfamide, Carboplatin, Etoposide, Bortezomib — Bortezomib starting at 1 mg/m(2), and escalating to 1.3, 1.5, 1.7. Bortezomib will be given on Days 1 (prior to rituximab) and 4, rituximab at 375 mg/m(2) on day 1, carboplatin AUC 5 and ifosfamide with mesna, each 5 mg/m(2), on day 3 and etoposide 100 mg/m(2)/day on days 2, 3, and 4 of a 21-day cycle. They will also receive filgrastim on days 6-13 or pegfilgrastim on day 6

SUMMARY:
This study seeks to determine the maximum tolerated dose of bortezomib in combination with rituximab, ifosfamide, carboplatin, and etoposide for patients with relapsed or primary refractory aggressive B-Cell Non-Hodgkin's lymphoma (diffuse large B-cell, mantle cell, follicular grade III, transformed lymphoma). Subjects will be enrolled in cohorts of 3 at each bortezomib dose level, starting at 1 mg/m(2), and escalating to 1.3, 1.5, and 1.7 mg/m(2). Bortezomib will be given on days 1 (prior to rituximab) and 4, rituximab 375 mg/m(2)/day on days 2, 3, and 4 of a 21-day cycle. They will also receive filgrastim on days 6-13 or pegfilgrastim on day 6.

ELIGIBILITY:
Inclusion Criteria:

* Aggressive B-Cell Lymphoma, CD-20 positive, in first relapse or refractory to first-line chemotherapy

  * Diffuse large B-cell Lymphoma, Mantle cell lymphoma, Follicular lymphoma (Grade III), Transformed Follicular Lymphoma
  * Rituximab is allowed
  * Prior radiation is allowed
* 18-70 years of age
* ECOG performance status of 0-2
* HIV seronegative
* Measurable disease on CT scan by international working group response criteria
* No CNS involvement
* Subject is considered to be a candidate for autologous stem cell transplant in the opinion of the treating physician
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control
* Male subject agrees to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Platelet count of <75 x 10(9)/L
* Absolute neutrophil count of <1.0 x 10(9)/L
* Calculated or measured creatinine clearance of <60 mL/minute within 14 days before enrollment
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Subject has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding.
* Subject has been treated with more than one prior chemotherapy regimen.
* Subject has received other investigational drugs with 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
-Determine the maximum tolerated dose of bortezomib in combination with rituximab, ifosfamide, carboplatin, and etoposide for patients with relapsed or primary refractory aggressive B-cell NHL | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D. Kaplan, M.D., Principal Investigator — University of California, San Francisco; Caroline Behler, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Cancer Center — http://cancer.ucsf.edu